CLINICAL TRIAL: NCT00916019
Title: Investigation on Gene Expression and Gene Marker Accompanied by a Single Bout of Exercise and Exercise Training
Brief Title: Investigation of the Effects of Exercise on Gene Expression
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fukuoka University (Other)
Responsible Party: Hiroaki Tanaka, Ph.D, Fukuoka University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 19200049
Record Dates: First submitted 2009-06-04; First posted 2009-06-08 (Estimated); Last update posted 2009-06-16 (Estimated); Status verified 2009-06

CONDITIONS: Healthy
Keywords: gene expression; skeletal muscle; Healthy men
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exercise (Experimental): mild exercise training
  Interventions: Other: exercise training

INTERVENTIONS:
Other: exercise training — 60 min of low-intensity exercise, 5 days/week, 12 weeks

SUMMARY:
The investigators have previously shown that mild exercise training at the level of lactate threshold (LT) intensity (60 min/day, 5 days/week) improves peripheral insulin sensitivity and insulin-independent glucose disposal of glucose effectiveness, without changes in body weight and body fat (Nishida et al, Diabetes Care, 2001; Nishida et al, Diabetes, 2004). Thus these beneficial effects are likely related to a number of adaptations that occur in skeletal muscle as response to exercise. In the current study, the investigators hypothesised that a single bout of mild exercise performed at LT would be a physiological stimulator of skeletal muscle PGC-1alpha gene, and the repetition of this exercise stimulating PGC-1alpha gene (i.e., training) for 12 weeks would induce coordinated increases in a large number of metabolic genes, as well as other genes potentially important in the prevention of insulin resistance and metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Men who were all in good health
* All individuals were free from diabetes and none were taking any medications
* All subjects were asked not to change their normal dietary habits, and not to engage in any strenuous physical activity

Exclusion Criteria:

* People who undergone regular exercise for at least 2 years
* Smokers

Ages: 19 Years to 32 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2002-07; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle PGC-1alpha gene expression and mitochondrial gene expression | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Hiroaki Tanaka, Ph.D., Principal Investigator — Fukuoka University
Locations (1):
- Fukuoka University, Fukuoka, Fukuoka, Japan